CLINICAL TRIAL: NCT02704000
Title: Home Visiting Programs to Improve Early Childhood Development and Maternal Mental Health - Evidence From the Western Region Cohort Project
Brief Title: Home Visiting Programs to Improve Early Childhood Development and Maternal Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Alexandra Brentani, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 38350114.0.0000.0076
Record Dates: First submitted 2016-02-24; First posted 2016-03-09 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Child Development; Mental Health Wellness 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No interventions - only baseline and endline assessments to be conducted at children's home.
- Home visits by CDAs (Experimental): Intervention: Behavioral: Home visiting program (Jamaica curriculum) Children in this intervention arm will be visited twice a months by trained child development agents (CDAs). CDAs will implement the Jamaica curriculum intervention during the home visits..
  Interventions: Behavioral: Home visiting program (Jamaica curriculum)
- Home visits by CHWs (Experimental): Intervention: Behavioral: Home visiting program (Jamaica curriculum) Children in this intervention arm will be visited twice a months by trained community health workers (CHWs) trained on delivering the intervention. CHWs will implement the Jamaica curriculum intervention during the home visits..
  Interventions: Behavioral: Home visiting program (Jamaica curriculum)

INTERVENTIONS:
Behavioral: Home visiting program (Jamaica curriculum) — Agents will deliver bi-weekly home-visits following the curriculum developed for the Jamaica intervention study by Susan Walker and colleagues. This curriculum foresees age-appropriate tasks assigned to the caregiver during each visit.
  Arms: Home visits by CDAs; Home visits by CHWs

SUMMARY:
This study evaluates the efficacy and cost-effectiveness of two platforms for delivering home visiting programs in the poor urban setting of Sao Paulo's western region: a program delivered by a newly trained cadre of Child Development Agents, and a program delivered by Community Health Agents employed by the government as part of the Family Health Strategy (ESF). The program will randomly select 400 mother-child dyads to follow a curriculum that is currently being adapted to the local context. The primary outcome of the program will be cognitive development for children aged 9 to 15 months old at baseline (21-27 months at endline) The secondary outcomes will include child physical development as well as maternal mental health.

DETAILED DESCRIPTION:
Despite major improvements in nutrition and child survival, a large share of children growing up in poor urban areas of Brazil continue to be exposed to a substantial amount of adversity in early childhood due to exposure to pollutants, exposure to external and domestic violence, unstable family environment, maternal depression and inadequate learning opportunities.

In this project we propose to assess the feasibility, impact and cost-effectiveness of home visiting programs in poor urban families living in Sao Paulo through a small-scale randomized pilot intervention accompanied by a rigorous impact evaluation. Home visiting programs do not only have the potential to improve maternal well-being, but have also been proven effective in increasing early life stimulation and child development.

Two delivery platforms for home visiting programs will be assessed as part of this trial: 1) the introduction of a newly trained cadre of Child Development Agents (CDAs); and 2) the integration of home visiting programs into the Family Health Strategy (PSF). For the latter, we will train selected Community Health Agents (CHA) currently employed by the Brazilian government under the Family Health Strategy program on child development and provide additional financial incentives for home visits. While this second option will be less costly, the quality of the delivered interventions may not be as high as the former. The developmental impact of both delivery mechanisms will be assessed. Impact data will be combined with detailed costing data to evaluate both the effectiveness and relatively cost-effectiveness of both platforms. Quantitative data on cost and developmental impact will be combined with qualitative feedback from mothers and community workers.The successful implementation of the pilot program may lead to a larger-scale efficacy and cost-effectiveness trial in Sao Paulo in the medium run, with the ultimate objective to establish similar programs at the national level in the long run.

Several recent studies from a wide range of countries such as Bangladesh, China, India Jamaica and South Africa have demonstrated that home visiting programs can be highly effective in improving child developmental outcomes.

The principal common feature of home visiting programs is that trained child development or community agents meet with mothers or parents on a regular basis to observe the interactions between caregivers and their children, and to provide practical guidance on how to interact with them. At the core of these visiting programs is a detailed curriculum, which contains key topics of child health and development to be covered at each home visit. Detailed information and supporting materials for each session have been developed for the original Jamaica study and are currently being adapted to the Brazilian context. In this project, we will assess the effectiveness and cost-effectiveness of the newly adapted home visiting programs in the poor urban context of Sao Paulo, Brazil. Given that Brazil's middle and upper income children already benefit from a range of early childhood care services, our focus will be low-SES families. Brazil currently offers a free health care system (SUS), which is primarily used by the low SES groups, according to the latest estimates 55.6 percent of urban households in Sao Paulo - these households will be the target population for the interventions, a group of 400 low SES mother-child dyads from Sao Paulo's western region.

The poor urban neighborhoods of São Paulo are representative of a large and rapidly growing group of urban settlements in low and middle-income countries. Many of these urban settings are - just like the household in the target area - not only characterized by exposure to a large variety of environmental hazards, but often also by high prevalence of domestic and external violence and lacking social support.

The target population of this project is low SES families from Sao Paulo's western region. As part of an ongoing research study (the Western Region Project), 6000 mother-child dyads have been enrolled in a longitudinal study, which means that detailed records on family background and birth outcomes will be available to this project. The second enabling factor is the tight integration of the research project into the larger health system, which will be beneficial for the recruitment and training of health workers and when it comes to connecting with families.

The main challenge faced by the project is the general lack of stability and trust in the targeted areas. Families residing in informal settlements, often illegal, tend to move frequently, and are often not willing to receive or interact with strangers. In some neighborhoods, outsiders are not welcome at all, so that regular meetings with mothers will be difficult. The strong links with the University Hospital should help overcome these barriers; local sensitization meetings will be organized to reduce the risk of refusals and attrition.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in Western Region Cohort study

Exclusion Criteria:

* not enrolled in Western Region Cohort study
* not in target age range

Ages: 9 Months to 17 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 826 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Child cognitive development as measured by Griffith Scales of Mental Development | 12 months after program initiation
  Overall cognitive development of children after 12 months of intervention.

SECONDARY OUTCOMES:
Maternal depression risk as assessed by the Edinburgh Scale | 12 months after program initiation
  The Edinburgh Scale assesses the risk of maternal depression
Child height relative to WHO reference curve (normalized z-score) | 12 months after program initiation
  Home measurement of children's height - scores will be normalized using WHO reference tables.
Child weight relative to WHO reference curve (normalized z-score) | 12 months after program initiation
  Home measurement of children's weight - weight in grams will be normalized using WHO reference tables.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra VM Brentani, PhD, Principal Investigator — Universidade de São Paulo, Faculdade de Medicina USP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brentani A, Walker S, Chang-Lopez S, Grisi S, Powell C, Fink G. A home visit-based early childhood stimulation programme in Brazil-a randomized controlled trial. Health Policy Plan. 2021 Apr 21;36(3):288-297. doi: 10.1093/heapol/czaa195. PMID 33496330
- [Result] Smith JA, Baker-Henningham H, Brentani A, Mugweni R, Walker SP. Implementation of Reach Up early childhood parenting program: acceptability, appropriateness, and feasibility in Brazil and Zimbabwe. Ann N Y Acad Sci. 2018 May;1419(1):120-140. doi: 10.1111/nyas.13678. PMID 29791729